CLINICAL TRIAL: NCT00302666
Title: Comparative, Prospective, Multi-Center, Open, Randomized Study to Investigate Bleeding Patterns, Metabolic Effects, Contraceptive Efficacy, Acceptance, and Safety of an Oral Contraceptive Containing 0.03 mg Ethinylestradiol and 2 mg Dienogest, in Two Different Regimens of Intake (Four Extended Cycles of 84 Days Each Versus the Conventional Regimen of 21 Days) in Healthy Volunteers
Brief Title: Bleeding Pattern Study
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Therapeutic Area Head, Bayer Schering Pharma AG
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 91227; 306903
Record Dates: First submitted 2006-02-23; First posted 2006-03-14 (Estimated); Last update posted 2009-05-18 (Estimated); Status verified 2009-05

CONDITIONS: Oral Contraceptive
Keywords: Contraception, Bleeding pattern

ARMS (2):
- Arm 1 (Sham Comparator)
  Interventions: Drug: Valette (Dienogest/EE30, BAY86-5038)
- Arm 2 (Sham Comparator)
  Interventions: Drug: Valette (Dienogest/EE30, BAY86-5038)

INTERVENTIONS:
Drug: Valette (Dienogest/EE30, BAY86-5038) — Oral contraceptive extended cycles
  Arms: Arm 1
Drug: Valette (Dienogest/EE30, BAY86-5038) — Oral contraceptive conventional cycles
  Arms: Arm 2

SUMMARY:
The aim of this study is to evaluate bleeding pattern, cycle control, contraceptive efficacy and safety of this oral contraceptive in two different regimens of intake.

DETAILED DESCRIPTION:
The study has previously been posted by Schering AG, Germany. Schering AG, Germany has been renamed to Bayer Schering Pharma AG, Germany.

Bayer Schering Pharma AG, Germany is the sponsor of the trial.

ELIGIBILITY:
Inclusion Criteria:

* Healthy female volunteers aged between 18 and 40 years requiring contraception.

Exclusion Criteria:

* Pregnancy or lactation.
* Any conditions that might interfere with the outcome as well as all contraindications for OC use.

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 1315 (Actual)
Dates: Start 2003-06; Study Completion 2005-02 (Actual)

PRIMARY OUTCOMES:
Bleeding pattern

SECONDARY OUTCOMES:
Safety, contraceptive efficacy

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (33):
- Germany (33):
  - Eberbach, Baden-Wurttemberg
  - Höchstadt A. D. Aisch, Bavaria
  - Krumbach, Bavaria
  - Neubiberg, Bavaria
  - Nuremberg, Bavaria
  - Hamburg, Hamburg
  - Dietzenbach, Hesse
  - Frankfurt am Main, Hesse
  - Fulda, Hesse
  - Kelkheim, Hesse
  - Langen, Hesse
  - Mühlheim am Main, Hesse
  - Hanover, Lower Saxony
  - Ronnenberg, Lower Saxony
  - Neustrelitz, Mecklenburg-Vorpommern
  - Gevelsberg, North Rhine-Westphalia
  - Gütersloh, North Rhine-Westphalia
  - Kirchheimbolanden, Rhineland-Palatinate
  - Speyer, Rhineland-Palatinate
  - Döbeln, Saxony
  - Dresden, Saxony
  - Leipzig, Saxony
  - Wurzen, Saxony
  - Bernburg, Saxony-Anhalt
  - Blankenburg, Saxony-Anhalt
  - Jessen, Saxony-Anhalt
  - Magdeburg, Saxony-Anhalt
  - Berlin, State of Berlin
  - Eisenberg, Thuringia
  - Gera, Thuringia
  - Jena, Thuringia
  - Kahla, Thuringia
  - Saalfeld, Thuringia